CLINICAL TRIAL: NCT07352566
Title: Utilization of a Cutaneous Therapy In Situ Microdevice
Brief Title: Utilization of a Microdevice for Psoriasis and Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 25-43621
Record Dates: First submitted 2025-11-17; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis; Atopic Dermatitis
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic | interventions — Triamcinolone; Fluorouracil; calcipotriene; tapinarof; crisaborole; Tacrolimus; Adalimumab; Etanercept; Certolizumab Pegol; Infliximab; secukinumab; ixekizumab; apremilast; risankizumab; Ustekinumab; Hydroxychloroquine; Methotrexate; Mycophenolic Acid; Azathioprine; Chloroquine; Cyclosporine; tofacitinib; deucravacitinib; dupilumab; tralokinumab; guselkumab; tildrakizumab; abrocitinib; upadacitinib; lebrikizumab; nemolizumab; ruxolitinib; bimekizumab; Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- In situ cutaneous microdevice (Experimental): The small device, about the size of a grain of rice, has up to 20 tiny reservoirs that hold medications that are approved by the Food and Drug Administration (FDA) for atopic dermatitis and psoriasis. Very small amounts of these medications will be released into the skin (at levels in your body much lower than are typically used). In this study, the device will be tested to see if it's safe and works well for predicting how the skin will react to standard treatments. We will also look at how these reactions are connected to genetic information and overall treatment results.
  Interventions: Device: In situ cutaneous microdevice; Drug: Triamcinolone; Drug: 5-Fluorouracil; Drug: Calcipotriene; Drug: Tapinarof; Drug: Crisaborole; Drug: Tacrolimus; Drug: Adalimumab; Drug: Etanercept; Drug: Certolizumab; Drug: Infliximab; Drug: Secukinumab; Drug: Ixekizumab; Drug: Apremilast; Drug: Risankizumab; Drug: Ustekinumab; Drug: Hydroxychloroquine; Drug: Methotrexate; Drug: Mycophenolate; Drug: Azathioprine; Drug: Chloroquine; Drug: Cyclosporine; Drug: Tofacitinib; Drug: Deucravacitinib; Drug: Dupilumab; Drug: Tralokinumab; Drug: Guselkumab; Drug: Tildrakizumab; Drug: Baractinib; Drug: Abrocitinib; Drug: Upadacitinib; Drug: Lebrikizumab; Drug: Nemolizumab; Drug: Ruxolitinib; Drug: Bimekizumab; Drug: Roflumilast

INTERVENTIONS:
Device: In situ cutaneous microdevice — The small device, about the size of a grain of rice, has up to 20 tiny reservoirs that hold medications that are approved by the Food and Drug Administration (FDA) for atopic dermatitis and psoriasis. In this study, the device will be tested to see if it's safe and works well for predicting how the skin will react to standard treatments. The microdevice will contain a subset of the following: Triamcinolone, 5-fluorouracil, Calcipotriene, Tapinarof, Crisaborole, Tacrolimus, Adalimumab, Etanercept, Certolizumab, Infliximab, Secukinumab, Ixekizumab, Apremilast, Risankizumab, Ustekinumab, Hydroxychloroquine, Methotrexate, Mycophenolate, Azathioprine, Chloroquine, Cyclosporine, Tofacitinib, Deucravacitinib, Dupilumab, Tralokinumab, Guselkumab, Tildrakizumab, Baractinib, Abrocitinib, Upadacitinib, Lebrikizumab, Nemolizumab, Ruxolitinib, Bimekizumab, Roflumilast.
Drug: Triamcinolone — Triamcinolone
Drug: 5-Fluorouracil — 5-fluorouracil
Drug: Calcipotriene — Calcipotriene
Drug: Tapinarof — Tapinarof
Drug: Crisaborole — Crisaborole
Drug: Tacrolimus — Tacrolimus
Drug: Adalimumab — Adalimumab
Drug: Etanercept — Etanercept
Drug: Certolizumab — Certolizumab
Drug: Infliximab — Infliximab
Drug: Secukinumab — Secukinumab
Drug: Ixekizumab — Ixekizumab
Drug: Apremilast — Apremilast
Drug: Risankizumab — Risankizumab
Drug: Ustekinumab — Ustekinumab
Drug: Hydroxychloroquine — Hydroxychloroquine
Drug: Methotrexate — Methotrexate
Drug: Mycophenolate — Mycophenolate
Drug: Azathioprine — Azathioprine
Drug: Chloroquine — Chloroquine
Drug: Cyclosporine — Cyclosporine
Drug: Tofacitinib — Tofacitinib
Drug: Deucravacitinib — Deucravacitinib
Drug: Dupilumab — Dupilumab
Drug: Tralokinumab — Tralokinumab
Drug: Guselkumab — Guselkumab
Drug: Tildrakizumab — Tildrakizumab
Drug: Baractinib — Baractinib
Drug: Abrocitinib — Abrocitinib
Drug: Upadacitinib — Upadacitinib
Drug: Lebrikizumab — Lebrikizumab
Drug: Nemolizumab — Nemolizumab
Drug: Ruxolitinib — Ruxolitinib
Drug: Bimekizumab — Bimekizumab
Drug: Roflumilast — Roflumilast

SUMMARY:
This study is being done to test a microdevice, which is a small device designed to test drugs directly on skin conditions like atopic dermatitis (eczema) and psoriasis.

The small device, about the size of a grain of rice, has up to 20 tiny reservoirs that hold medications that are approved by the Food and Drug Administration (FDA) for atopic dermatitis and psoriasis. Very small amounts of these medications will be released into the skin (at levels in your body much lower than are typically used). In this study, the device will be tested to see if it's safe and works well for predicting how the skin will react to standard treatments. We will also look at how these reactions are connected to genetic information and overall treatment results.

ELIGIBILITY:
Inclusion Criteria:

> 18 years of age patients with atopic dermatitis or psoriasis if female patient with child bearing potential (on oral contraceptive pills or intrauterine device for at least 30 days)

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 1 year
  The safety of microdevice placement and removal will be based on assessment of adverse events.
Proportion of retrieved devices with assessable tissue | 1 year
  The feasibility of microdevice analysis based on the ability to place and retrieve the device with sufficient tissue, of sufficient quality, for downstream histopathology/molecular analysis and interpretation of at least 80% of the device reservoirs.

SECONDARY OUTCOMES:
Change in local skin inflammation (molecular assays) | 1 year
  Feasibility of utilizing quantitative histopathologic assessment and/or transcriptional profiling to determine whether there is local change in lesional rash-affected skin with clinically relevant skin inflammation treating agents.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Cho, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsai LL, Phillips WW, Hung YP, Dominas C, Deans K, Ahn S, Ferland B, Weiss K, Lanuti M, Auchincloss H, Schumacher L, Jonas O, Colson YL. First-in-Human Intrathoracic Implantation of Multidrug-Eluting Microdevices for In Situ Chemotherapeutic Sensitivity Testing as Proof of Concept in Nonsmall Cell Lung Cancer. Ann Surg. 2023 May 1;277(5):e1143-e1149. doi: 10.1097/SLA.0000000000005385. Epub 2023 Apr 6. PMID 35129472
- [Background] Tatarova Z, Blumberg DC, Korkola JE, Heiser LM, Muschler JL, Schedin PJ, Ahn SW, Mills GB, Coussens LM, Jonas O, Gray JW. A multiplex implantable microdevice assay identifies synergistic combinations of cancer immunotherapies and conventional drugs. Nat Biotechnol. 2022 Dec;40(12):1823-1833. doi: 10.1038/s41587-022-01379-y. Epub 2022 Jul 4. PMID 35788566
- [Background] Peruzzi P, Dominas C, Fell G, Bernstock JD, Blitz S, Mazzetti D, Zdioruk M, Dawood HY, Triggs DV, Ahn SW, Bhagavatula SK, Davidson SM, Tatarova Z, Pannell M, Truman K, Ball A, Gold MP, Pister V, Fraenkel E, Chiocca EA, Ligon KL, Wen PY, Jonas O. Intratumoral drug-releasing microdevices allow in situ high-throughput pharmaco phenotyping in patients with gliomas. Sci Transl Med. 2023 Sep 6;15(712):eadi0069. doi: 10.1126/scitranslmed.adi0069. Epub 2023 Sep 6. PMID 37672566
- [Background] Jonas O, Landry HM, Fuller JE, Santini JT Jr, Baselga J, Tepper RI, Cima MJ, Langer R. An implantable microdevice to perform high-throughput in vivo drug sensitivity testing in tumors. Sci Transl Med. 2015 Apr 22;7(284):284ra57. doi: 10.1126/scitranslmed.3010564. PMID 25904741

DOCUMENTS (2):
  • Study Protocol (2025-11-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT07352566/Prot_000.pdf
  • Statistical Analysis Plan (2025-11-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT07352566/SAP_001.pdf